CLINICAL TRIAL: NCT07221305
Title: Feasibility and Efficacy of Delivering a Mobile Application-Based Neuromuscular Training Program to High School Athletes: Adherence, Agility, and Single Leg Squat Kinematics
Brief Title: RIIP REPS Neuromuscular Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB #2023-0499
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Neuromuscular Control; Healthy; Athletic Performance and Injury Risk
Keywords: Neuromuscular Control Training; Injury Prevention; High School Athletes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuromuscular Control Training Program (Experimental): The intervention was a self-paced neuromuscular control training program that athletes completed on their mobile phones via the RIIP REPS app. Athletes were instructed to complete 4 sessions per week throughout the 6 week intervention.
  Interventions: Other: Neuromuscular Control Training

INTERVENTIONS:
Other: Neuromuscular Control Training — The mobile app-based neuromuscular control training program was administered via the RIIP REPS application. The program consisted of 24 unique 7-minute sessions. Each session emphasized bodyweight training targeting landing mechanics, trunk and hip control, balance, and posterior chain engagement. The sessions progressed in difficulty throughout the intervention.
  Other Names: Neuromuscular Training; NMT

SUMMARY:
The purpose of this study is to assess both the feasibility and efficacy of a 6-week mobile-application-based neuromuscular training program in high school athletes by measuring adherence rates and examining changes in agility and neuromuscular control. Outcomes were measured both during the intervention (adherence) as well as at pre- and post-intervention data collection sessions.

DETAILED DESCRIPTION:
This study recruited high school athletes (ages 14-18) from Westchester County, NY to participate in a six week mobile application-based neuromuscular control training program that was downloaded onto each participant's personal smartphone and consisted of 24 unique 7-minute sessions. Pre/post intervention assessments included (1) an agility T test and (2) a video-recorded single leg squat test from sagittal and coronal planes. Sagittal plane analysis captured peak knee and hip flexion angles; coronal plane analysis assessed alignment of the knee, hips, and trunk. These subcomponent scores were combined into an 8-point composite movement quality score previously described by Di Paolo et al. Paired t-tests and effect sizes (Cohen's d) were computed to evaluate pre-post changes in agility T test performance and Di Paolo single leg squat composite and subcomponent scores. Participants were arranged by adherence into high (≥12 sessions) and low (<12 sessions) groups to determine if any relationship existed between adherence and outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-18
* Actively participating in an organized sport OR have participated in an organized sport in the last 12 months
* Pre-intervention testing completed AND post-intervention testing completed within 2 weeks of completing the 6 week program

Exclusion Criteria:

* Individuals whose physical activity and/or sports participation is currently limited by an illness or injury
* Individuals with previous lower extremity injury and/or surgery
* Individuals who are not fluent in English
* Individuals without access to an iOS or Android mobile phone

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Compliance | Throughout the 6 week intervention
  Compliance with the RIIP REPS mobile program was defined by how many sessions were completed by each participant. Full compliance consisted of the recommended four sessions per week for a total of 24 sessions over the 6 week period. Adherence tiers were determined based on the number of sessions completed and were as follows: low adherence (<12 sessions), and high adherence (>12 sessions).

SECONDARY OUTCOMES:
Movement Quality | Testing was performed before and within 2 weeks after the 6 week intervention.
  Athletes completed a total of 12 single-leg squats (SLS), guided by trained sports medicine educators. The test protocol consisted of three SLS per leg in the frontal plane and three in the sagittal plane. In the frontal plane, the athlete faced the camera; for the sagittal plane, the athlete turned 90 degrees, maintaining the same squatting leg toward the camera. If a participant lost balance during a repetition, they were instructed to repeat the squat to ensure three successful trials per view. Videos were then analyzed based on the criteria set forth by Di Paolo et al. and the measurements were then used to compute a composite score (0 through 8) with a higher score indicating better performance.
Agility T Test | Testing was performed before and within 2 weeks after the 6 week intervention.
  The T test is a widely used measure of change-of-direction speed and agility, consisting of a T-shaped running course that challenges lateral, forward, and backward movement. Athletes began at the base of the "T," sprinted forward 10 yards to touch a central cone, shuffled 5 yards to one side to touch another cone, shuffled 10 yards laterally to the opposite side to touch a second cone, returned to the center cone via shuffle, and then backpedaled to the starting point. Proper technique and cone touches were required for a valid trial. To ensure timing accuracy, each trial was independently timed by two study personnel using handheld stopwatches. The average of the two recorded times was used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Pearle, M.D., Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petushek EJ, Sugimoto D, Stoolmiller M, Smith G, Myer GD. Evidence-Based Best-Practice Guidelines for Preventing Anterior Cruciate Ligament Injuries in Young Female Athletes: A Systematic Review and Meta-analysis. Am J Sports Med. 2019 Jun;47(7):1744-1753. doi: 10.1177/0363546518782460. Epub 2018 Jul 12. PMID 30001501
- [Background] Steib S, Rahlf AL, Pfeifer K, Zech A. Dose-Response Relationship of Neuromuscular Training for Injury Prevention in Youth Athletes: A Meta-Analysis. Front Physiol. 2017 Nov 14;8:920. doi: 10.3389/fphys.2017.00920. eCollection 2017. PMID 29184511
- [Background] Di Paolo S, Musa F, d'Orsi GM, Grassi A, Vulpiani MC, Zaffagnini S, Della Villa F. A comprehensive two-dimensional scoring system to assess the single-leg squat task in football players. Knee. 2024 Jun;48:52-62. doi: 10.1016/j.knee.2024.02.016. Epub 2024 Mar 20. PMID 38513322